CLINICAL TRIAL: NCT01767454
Title: Phase 1 Study of the BRAF Inhibitor Dabrafenib +/- MEK Inhibitor Trametinib in Combination With Ipilimumab for Unresectable or Metastatic Melanoma
Brief Title: Study of Dabrafenib +/- Trametinib in Combination With Ipilimumab for V600E/K Mutation Positive Metastatic or Unresectable Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115984
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumours
Keywords: BRAF V600E; Melanoma; V600K; Trametinib; Dabrafenib; Ipilimumab
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doublet arm (Experimental): Subjects will be started with dabrafenib 150 mg twice daily (BID) orally for 2 weeks (run-in). The doublet arm will comprise 2 cohorts. Cohort A1 (Dabrafenib 150 mg BID + ipilimumab). Cohort A-1 (Dabrafenib 100 mg BID +ipilimumab). Ipilimumab will be administered as 3 mg/kg every 3 weeks (Q3W) for a total of 4 infusions over approximately 12-16 weeks. Dabrafenib will be continued through combination with ipilimumab and post-ipilimumab until no longer of clinical benefit, in the opinion of the treating physician, or until unacceptable AE or death
  Interventions: Drug: Dabrafenib; Drug: Ipilimumab
- Triplet arm (Experimental): This arm will be initiated using dabrafenib and ipilimumab doses established in the doublet dose-finding. Subjects will be started with dabrafenib and trametinib orally for 2 weeks (run-in), followed by ipilimumab 3 mg/kg Q3W for a total of 4 infusions over approximately 12-16 weeks. The triplet arm will comprise 3 planned cohorts. Cohort B-1: Dabrafenib 100 mg BID + trametinib 1 mg once daily + ipilimumab, Cohort B1: Dabrafenib 150 mg BID + trametinib 1 mg once daily+ ipilimumab, Cohort B2: Dabrafenib 150 mg BID + trametinib 2 mg once daily + ipilimumab. Dabrafenib and trametinib wil be continued through combination with ipilimumab and post-ipilimumab until no longer of clinical benefit, in the opinion of the treating physician, or until unacceptable AE or death
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Ipilimumab

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib 100 mg or 150 mg BID orally will be administered. Capsules with unit dose strengths of 50 mg or 75 mg
Drug: Trametinib — Trametinib 1 mg or 2 mg once daily will be administered. Tablets with unit dose strengths of 0.5 mg or 2 mg
  Arms: Triplet arm
Drug: Ipilimumab — Ipilimumab 3 mg/kg intravenously over 90 minutes Q3W for a total of 4 doses will be administered. Supplied as Vials of 50 mg/10 mL (5 mg/mL) and 200 mg/40 mL (5 mg/mL)

SUMMARY:
This is an open-label, multi-center, dose-finding Phase 1 study that will enroll subjects at least 18 years old with unresectable or metastatic melanoma and BRAF V600 mutations. The primary objective of the study is to describe the safety for the doublet therapy (dabrafenib and ipilimumab) and the triplet therapy (dabrafenib/trametinib and ipilimumab). Preliminary efficacy data will also be collected. Subjects will be assigned to receive either the doublet combination (dabrafenib and ipilimumab) or the triplet combination (dabrafenib, trametinib, and ipilimumab). Subjects will be enrolled to dose-finding cohorts in the doublet combination (dabrafenib + ipilimumab) in a sequential 3+3 fashion. Following establishment of a dose for the doublet combination, an expansion cohort will be opened. At the same time, enrollment to dose finding cohorts for the triplet combination (dabrafenib + trametinib + ipilimumab) will begin in a sequential 6+6 fashion. Enrollment into triplet cohorts will take priority when both the doublet expansion arm and the triplet dose-finding arm are open for enrollment at the same time. Approximately 9-24 subjects will be enrolled to the dose finding portion of the study. Approximately 30 subjects will be enrolled to doublet expansion cohort and 30 subjects will be enrolled in the triplet expansion cohort. A two-week run-in period without ipilimumab will be followed by 4 intravenous doses of ipilimumab at the recommended dose and schedule. Oral daily dosing of dabrafenib or dabrafenib + trametinib will continue from the two-week run-in, through combination with ipilimumab, and post-ipilimumab until no longer of clinical benefit, in the opinion of the treating physician, or until unacceptable AE or death

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Males and females >= 18 years of age
* Histologically confirmed cutaneous melanoma that is either Stage IIIc (unresectable) or Stage IV (metastatic), and determined to be BRAF V600E or V600K mutation-positive by the local laboratory. Subjects with ocular or mucosal melanoma are not eligible
* Measurable tumor by physical or radiographic examination
* Subjects must not have had more than 1 previous treatment regimen with chemotherapy, interferon, or IL-2 for metastatic melanoma
* All prior anti-cancer treatment-related toxicities (except alopecia) must be <= Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 at the time of enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate baseline organ function as defined by: absolute neutrophil count (ANC) >= 1.2 × 109/L; Hemoglobin >= 9 g/dL; Platelet count >= 100 x 109/L; prothrombin time (PT) / international normalized ratio (INR) and partial thromboplastin time (PTT) <= 1.5 x upper limit of normal (ULN); Albumin >= 2.5 g/dL; Total bilirubin <= 1.5 x ULN; aspartate aminotransferase (AST) and alanine transaminase (ALT) <= 2.0 x ULN; Creatinine <=1.5 mg/mL; Left Ventricular Ejection fraction (LVEF) >= lower limit of normal (LLN) by ECHO
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization and agree to use effective contraception, during the study, and for 30 days after the last dose of study treatment
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception for at least 2 weeks prior to the first dose of study treatment until 16 weeks after the last dose of study treatment to allow for clearance of any altered sperm
* Able to swallow and retain orally administered study treatment and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels

Exclusion Criteria:

* Prior treatment with a BRAF inhibitor (including but not limited to dabrafenib, vemurafenib, and XL281/BMS-908662) or a MEK inhibitor (including but not limited to trametinib, AZD6244, and RDEA119) or ipilimumab or any other agent targeting a T-cell immunomodulatory pathway (including, but not limited to CTLA-4, PD-1, 4-1BB, OX40, GITR, CD27, and CD28)
* Any major surgery, extensive radiotherapy, chemotherapy with delayed toxicity, biologic therapy, or immunotherapy within 21 days prior to randomization and/or daily or weekly chemotherapy without the potential for delayed toxicity within 14 days prior to randomization
* Known Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection)
* A history of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Brain metastasis are excluded unless

  1. All known lesions were previously treated with surgery or stereotactic surgery (whole-brain radiation is not allowed unless given after definitive treatment with surgery or stereotactic surgery) AND
  2. Brain lesion(s), if still present, must be confirmed stable (i.e., no increase in lesion size) for >= 6 weeks prior to randomization (stability must be confirmed with two consecutive magnetic resonance image (MRI) or computed tomography (CT) scans with contrast, AND
  3. Asymptomatic with no corticosteroid requirements for >= 4 weeks prior to randomization, AND
  4. No enzyme inducing anticonvulsants for >= 4 weeks prior to randomization
* A history or evidence of cardiovascular risk including any of the following

  1. LVEF < LLN for the institution
  2. A corrected QT interval >=480 msec (e.g. Bazett's formula [QTcB])
  3. A history or evidence of current clinically significant uncontrolled arrhythmias (exception: subjects with controlled atrial fibrillation for > 30 days prior to randomization are eligible)
  4. A history (within 6 months prior to first dose of study treatment) of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty
  5. A history or evidence of current >=Class II congestive heart failure as defined by the New York Heart Association (NYHA)
  6. Treatment refractory hypertension defined as systolic blood pressure >140 millimetres of mercury (mmHg) and/or diastolic blood pressure >90 mmHg which cannot be controlled by antihypertensive therapy
  7. Patients with intra-cardiac defibrillators
  8. Abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study
* A history or current evidence/risk of retinal vein occlusion (RVO) or Central serous retinopathy (CSR) including

  1. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes), or
  2. Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR such as evidence of new optic disc cupping; Evidence of new visual field defects on automated perimetry; Intraocular pressure >21 mmHg as measured by tonography
* History of any of the following diseases: inflammatory bowel disease or any other autoimmune bowel disease; systemic lupus erythematosus; rheumatoid arthritis; or any autoimmune ocular diseases. Patients with active autoimmune disease or a history of autoimmune disease other than those mentioned above must be approved by the GSK medical monitor
* Active pneumonitis or interstitial lung disease
* Lactating female
* History of another malignancy (Exception: Subjects who have been disease-free for 3 years, or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible)
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures
* Any prohibited medication
* Administration of an investigational study treatment within 28 days or 5 half-lives, whichever is longer, preceding the first dose of study treatment(s) in this study
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO)
* Unwillingness or inability to follow the procedures outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-02-12 (Actual); Primary Completion 2015-09-04 (Actual); Study Completion 2015-09-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events (AEs) to assess the safety of dabrafenib +/- trametinib when administered in combination with ipilimumab | Follow-up up to 6 months after last subject last dose
  AEs will be collected from the time the first dose of study treatment is administered until 30 days following discontinuation of study treatment
Changes in laboratory values, vital signs, and physical examinations as a measure of safety of dabrafenib +/- trametinib when administered in combination with ipilimumab | Follow-up up to 6 months after last subject last dose
  Hematology, clinical chemistry, and urinalysis parameters to be tested. Vital sign measurements will include systolic and diastolic blood pressure, temperature, respiration rate and pulse rate. A complete physical examination will be performed at screening and every 12 months thereafter, as well as whenever clinically indicated.A brief physical examination will be performed every 3 or 4 weeks

SECONDARY OUTCOMES:
Number of subjects with AEs and changes in laboratory values, vital signs, and physical examinations to determine a recommended dose for dabrafenib +/- trametinib when administered in combination with ipilimumab | Up to approximately Week 9 in doublet and triplet arm
  All subjects will be evaluated for dose-limiting toxicity (DLT) from the first dose of ipilimumab until 1 week after the third dose of ipilimumab to determine a recommended dose for dabrafenib +/- trametinib when administered in combination with ipilimumab
Overall response rate | Follow-up up to 6 months after last subject last dose
  Overall Response will be determined using Modified immune-related response criteria (irRC)
Concentrations of trametinib, dabrafenib and its metabolites (GSK2285403, GSK2298683, and GSK2167542) in the triplet arm and dabrafenib and its metabolites in the doublet arm | Day 15 (pre-dose,1, 2, and 4 hours post-dose); Day 36 and Day 57 (pre-dose only) for doublet and triplet arms
  Four blood samples will be collected on the day of first dose of ipilimumab (Cycle 1) - Study Day 15. One blood sample will be obtained on the day of the second and third dose of ipilimumab (Cycles 2 and 3) - Study Days 36 and 57. Subjects will be instructed to withhold their morning dose until after they arrive at the clinic. Ipilimumab infusion should start as soon as possible after oral dosing of dabrafenib/trametinib. PK samples have a +/-30 minute window for collection.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Ackerman A, Klein O, McDermott DF, Wang W, Ibrahim N, Lawrence DP, Gunturi A, Flaherty KT, Hodi FS, Kefford R, Menzies AM, Atkins MB, Long GV, Sullivan RJ. Outcomes of patients with metastatic melanoma treated with immunotherapy prior to or after BRAF inhibitors. Cancer. 2014 Jun 1;120(11):1695-701. doi: 10.1002/cncr.28620. Epub 2014 Feb 27. PMID 24577748
- See also: Results for study BRF115984 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/115984?search=study&study_ids=BRF115984#rs